CLINICAL TRIAL: NCT02586610
Title: A Phase II Trial of Neoadjuvant Chemoradiation (CRT) and Pembrolizumab in Patients With Rectal Cancer: Hoosier Cancer Research Network GI15-213
Brief Title: Trial of Chemoradiation and Pembrolizumab in Patients With Rectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dr. Rahma decided to run the study through a different group
Sponsor: Osama Rahma, MD (Other)
Collaborators: Hoosier Cancer Research Network (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Osama Rahma, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GI15-213
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Rectal Cancer; Rectal Neoplasm
Keywords: Pembrolizumab; Chemoradiation; Anti-PD-1 Antibody; MK-3475
MeSH Terms: conditions — Rectal Neoplasms | interventions — pembrolizumab; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant Treatment (Experimental): All subjects will receive concurrent chemoradiation and pembrolizumab neoadjuvant treatment for 6 weeks:
  * Pembrolizumab 200 mg IV Days 1, 22 and 43
  * Capecitabine 825 mg/m2 PO in twice daily doses (total 1650 mg/m2) on 5 consecutive days / week M-F given on the radiation days for 28 days
  * Radiation therapy 50.4 GY. Daily fractions of 1.8 Gy over a 6 week interval, excludes weekends
  Interventions: Drug: Pembrolizumab; Drug: Capecitabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV Days 1, 22 and 43
  Other Names: MK-3475
Drug: Capecitabine — Capecitabine 825 mg/m2 PO twice a day (daily total 1650 mg/m2) on 5 consecutive days / week M-F given on the radiation days for 28 days
  Other Names: Xeloda
Radiation: Radiation Therapy — Radiation 50.4 GY in daily fractions of 1.8 Gy over a 6 week interval (excludes weekends)
  Other Names: XRT

SUMMARY:
This is a phase II, prospective open label multi-center study in which subjects with stage II-III rectal cancer will be accrued in order to determine the pathological complete response rate of neoadjuvant pembrolizumab in combination with chemoradiation treatment (CRT). Subjects must have a diagnosis of rectal cancer, stage II (T3-4, N0) or stage III (any T, N1-2). Subjects must have received no prior treatments (chemotherapy, pelvic radiation or surgery) for their rectal cancer.

Eligible subjects will receive standard chemoradiation with pembrolizumab administered every 3 weeks on days 1, 22, and 43 of the neoadjuvant interval. In all subjects, restaging endorectal or pelvic MRI with chest and abdominal CT will be performed at 6-8 weeks after completion of neoadjuvant treatment to determine resectability and to rule out any evidence of metastases. Subjects who have resectable disease will undergo surgery within 2-4 weeks of imaging; 8-12 weeks after completion of chemoradiation. Subjects who are found to have unresectable or metastatic disease post treatment with the combination of CRT+ pembrolizumab should receive standard of care definitive treatment per the discretion of their treating physician.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

NEOADJUVANT TREATMENT:

All subjects will receive concurrent chemoradiation and pembrolizumab neoadjuvant treatment for 6 weeks:

* Pembrolizumab 200 mg Intravenously (IV) Days 1, 22 and 43
* Capecitabine 825 mg/m2 PO (by mouth) in twice daily doses (daily total 1650 mg/m2) on 5 consecutive days / week Monday-Friday given on the radiation days for 28 days
* Radiation 50.4 Gy (Gray) in daily fractions of 1.8 Gy over a 6 week interval,excludes weekends

POST NEOADJUVANT TREATMENT:

* End of treatment (EOT) 6-8 weeks after last dose of neoadjuvant treatment, all subjects will be assessed to determine resectability. Those with resectable disease will undergo surgery within 2-4 weeks of imaging, 8-12 weeks after completion of chemoradiation. Subjects who are found to have unresectable or metastatic disease post treatment with the combination of CRT+ pembrolizumab should receive standard of care definitive treatment per the discretion of their treating physician.
* Surgical Resection ( 2-4 weeks after restaging imaging and 8-12 weeks after completion of chemoradiation)
* Follow Up
* Post Operative Visit (4-6 weeks after surgery)
* Disease Follow Up -Years 1-2 (per site investigator discretion; suggested every 3-6 months)
* Survival Follow Up - Years 3-5

To demonstrate adequate organ function, all screening labs should be performed within 7 days of treatment initiation:

Hematological:

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL
* Hemoglobin ≥9 g/dL without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)

Renal:

* Serum creatinine ≤1.5 X upper limit of normal (ULN) OR
* Measured or calculated creatinine clearance ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl

Hepatic:

* Serum total bilirubin ≤ 1.5 X ULN
* Aspartate transaminase (AST) / Serum glutamic oxaloacetic transaminase (SGOT) ≤ 2.5 X ULN
* Alanine aminotransferase (ALT) / Serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 X ULN
* Albumin ≥2.5 mg/dL

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants)

ELIGIBILITY:
Diagnosis/Condition for Entry into the Trial:

* Histologically confirmed adenocarcinoma of the rectum

  * Clinical stage II (T3-4, N-) or stage III (any T, N+) rectal cancer based on pelvic MRI.
  * Tumor located within 12 cm of the anal verge (determined by rigid proctoscopy or flexible sigmoidoscopy).

Subject Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be 18 years of age or older on day of signing informed consent.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1).
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
* Have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study treatment.

Subject Exclusion Criteria:

* Unresectable disease, as evidenced by invading adjacent organs and surgical resection will not achieve negative margins
* Recurrent rectal cancer
* Evidence of metastatic disease (as determined by chest and abdominal CT).
* Prior malignancy within the prior 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Prior radiation for other diagnoses to the expected rectal cancer treatment fields.
* Prior surgery, radiation, chemotherapy, targeted therapy, or investigational therapy for rectal cancer. NOTE: If subject received major surgery for reason other than rectal cancer, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the planned start of study treatment.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Administration of live vaccine within 30 days of planned start of study therapy. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Serious uncontrolled medical disorder that in the opinion of the site investigator would impair the ability of the subject to receive protocol therapy.
* Unable or unwilling to participate a study related procedure, including MRI.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Time from start of neoadjuvant chemoradiation until surgical resection (estimate up to 12 weeks after completion of chemoradiation)
  Proportion of subjects with pathological complete response (pCR) as demonstrated by the absence of residual invasive cancer on evaluation of the complete resected rectal specimen.

SECONDARY OUTCOMES:
Density of CD8(+) Tumor-Infiltrating Lymphocytes (TIL) | Time from baseline until completion of post-neoadjuvant treatment (estimate up to 8 weeks after completion of chemoradiation)
  Estimate the density of CD8 TILs in the tumor at baseline and post-neoadjuvant treatment
Response Rate (RR) | Time from registration to documented progression or subject death from any cause, assessed up to 42 months
  RR of subjects treated with the combination of chemoradiation and pembrolizumab, assessed using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) criteria.
Disease Free Survival (DFS) | Time from start of protocol treatment to the date of progression or death from any cause, whichever occurs first, assessed up to 42 months
  DFS of subjects treated with the combination of chemoradiation and pembrolizumab, assessed using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) criteria.
Overall Survival (OS) | Time from start of protocol treatment to death from any cause, assessed up to 42 months
  OS outcomes assessed using Kaplan-Meier Survival Analysis Subjects who have not died while on study or are lost to follow up will be censored at their last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Rahma, Study Chair — Hoosier Cancer Research Network

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org